CLINICAL TRIAL: NCT07381985
Title: Strategy for Management of Patients With Hereditary Cancer Syndromes (HCS) in a Rural Environment
Acronym: LINC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Kara Landry, Assistant Professor of Oncology & Hematology, University of Vermont Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00002507/UVMCC2204
Record Dates: First submitted 2025-05-08; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Cancer Syndromes; BRCA1 Hereditary Breast and Ovarian Cancer Syndrome; Lynch Syndrome
Keywords: Hereditary Cancer Syndromes; Lynch Syndrome; Rural Health
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Longitudinal Cancer Genetics Follow-Up Program (Experimental): Participants in this arm will be enrolled in a longitudinal cancer genetics follow-up program designed for individuals with known hereditary cancer syndromes (HCS). The intervention includes scheduled clinical visits with a cancer genetics physician and, as needed, a genetic counselor at baseline, 12 months, and 24 months. Participants will receive individualized care plans summarizing surveillance and prevention recommendations. Adherence, distress (MICRA), and care coordination (CCI) will be assessed through surveys administered at each visit.
  Interventions: Behavioral: Longitudinal Cancer Genetics Follow-Up Program

INTERVENTIONS:
Behavioral: Longitudinal Cancer Genetics Follow-Up Program — Participants will be enrolled in a structured, two-year longitudinal follow-up program designed for individuals with known hereditary cancer syndromes (HCS). The program includes baseline, 12-month, and 24-month clinic visits with a cancer genetics physician and, as needed, a genetic counselor. During each visit, participants will receive a personalized care plan outlining guideline-based cancer prevention and surveillance recommendations. Participants will also complete adherence surveys with their provider, and independently complete the MICRA and Care Coordination Index (CCI) surveys to assess distress and care coordination. Visits may be conducted in person or via televideo, based on clinical need and participant preference.

SUMMARY:
This study aims to improve cancer prevention and surveillance adherence in patients with Hereditary Cancer Syndromes (HCS), particularly those living in rural areas. The study will evaluate whether enrolling HCS patients in a longitudinal clinical program with individualized care plans and regular follow-up improves adherence to guideline-recommended cancer screening and risk-reduction strategies. Secondary aims include assessing the program's impact on patient distress and perceived care coordination. The study will enroll 200 adults with known pathogenic germline mutations who were previously seen at the UVM Medical Center genetics clinic. Participants will complete surveys at baseline, 12, and 24 months to assess adherence, distress, and care coordination. Findings from this study will inform future efforts to reduce gaps in hereditary cancer care delivery, especially for rural populations.

DETAILED DESCRIPTION:
This single-arm, prospective, interventional study will assess the feasibility and impact of a structured longitudinal follow-up program for patients with Hereditary Cancer Syndromes (HCS). Eligible participants will have a known pathogenic germline variant in a cancer risk gene identified by a CLIA-approved lab at least one year prior to enrollment. All participants will be seen at baseline and followed clinically for two years, with additional visits as clinically indicated. Each participant will receive an individualized care plan developed by cancer genetics providers and supported by annual follow-up visits.

The primary objective is to assess whether participation in this program increases adherence to National Comprehensive Cancer Network (NCCN) guideline-recommended cancer screening and prevention strategies (e.g., surveillance imaging, colonoscopy, prophylactic surgery). Secondary objectives include evaluating changes in participant distress and perceived care coordination over time, and examining how rurality (defined using RUCA codes) affects outcomes.

Participants will complete three study instruments at baseline, 12-month, and 24-month follow-up visits:

A gene-specific adherence survey administered by the genetics team,

The Multidimensional Impact of Cancer Risk Assessment (MICRA) questionnaire to assess distress,

The Care Coordination Index (CCI) to evaluate patient-perceived coordination of care.

A retrospective chart review of previously seen HCS patients will also be conducted to estimate baseline adherence rates and support feasibility assessments. Statistical analyses will use generalized probit and linear models to evaluate changes over time and assess effect modification by demographic and clinical variables such as age, sex, gene mutation, and rurality.

This study will generate critical pilot data to inform future controlled studies and improve access to high-quality cancer prevention care, particularly for underserved rural populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all genders must be ≥ 18 years of age.
* Patients must have a known pathogenic germline variant in a cancer risk gene that was identified by a CLIA-approved lab more than one year ago.
* Patients must be able to accurately provide self-report data (i.e., per clinical judgment, cognitive function is intact).
* Patients must be able to complete questionnaires in English.
* Patients must have the ability to provide informed consent.

Exclusion Criteria:

- Patients who tested positive for a germline pathogenic variant associated with cancer risk < 1 year ago are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to Cancer Prevention and Surveillance Guidelines | Baseline, 12 months, and 24 months
  Proportion of participants who are adherent to National Comprehensive Cancer Network (NCCN) guideline-recommended cancer risk-reducing strategies-including surveillance imaging, colonoscopy, chemoprevention, and prophylactic surgeries-measured at baseline, 12 months, and 24 months. Adherence will be determined through a gene-specific adherence survey completed during clinic visits and supported by clinical documentation.

SECONDARY OUTCOMES:
Change in Participant Distress Level as Measured by the MICRA Questionnaire | 2 years
  This outcome will assess change in participant distress related to hereditary cancer risk using the validated Multidimensional Impact of Cancer Risk Assessment (MICRA) questionnaire. The MICRA provides a total distress score and subscale scores for positive experiences, intrusive thoughts, and distress. Participants complete the MICRA at baseline, 12-month, and 24-month follow-up visits. Scores will be compared over time to evaluate the impact of enrollment in a longitudinal cancer genetics program on emotional distress. Unit of Measure:
  Mean change in MICRA total distress score.
Change in Perceived Care Coordination | 2 years
  This outcome will assess change in participants' perceived care coordination over time using the validated Care Coordination Index (CCI). The CCI is a participant-reported measure that evaluates multiple domains of care coordination. Scores range from 0 to 100, with higher scores indicating better perceived care coordination. Participants will complete the CCI at baseline, 12-month, and 24-month follow-up visits. Changes in scores will be analyzed to determine whether enrollment in a formal longitudinal follow-up program improves care integration.
  Unit of Measure: Mean change in Care Coordination Index (CCI) score
  Assessment Tool: Care Coordination Index (CCI) - participant-reported questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized patient related data will be incorporated into publications and will be made available to other investigators at reasonable request.